CLINICAL TRIAL: NCT00316056
Title: Using Virtual Reality to Test Communication Strategies for Genomic Concepts
Brief Title: Use of Virtual Reality to Communicate Concepts of Genomics to the General Public
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060143; 06-HG-0143
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-25

CONDITIONS: Healthy; Learning; Communication
Keywords: Genetic Literacy; Learning; Genetic Knowledge; Public Understanding of Science; Science Education; Healthy Volunteer; HV
MeSH Terms: conditions — Communication

SUMMARY:
This study will investigate how people learn best about genetics. It involves participating in activities in NHGRI's Immersive Virtual Environment Laboratory (IVE lab), where digital "virtual worlds" are created that appear to surround the subject when he or she wears a head-mounted display.

English-speaking men and women between 18 and 40 years of age may be eligible for this study. Participants are randomly assigned to one of two groups, each of which receives a different type of information, once in the IVE lab. Subjects complete a questionnaire before and after performing the activities in the lab. The questionnaire evaluates the subject's knowledge of genetics and tests some reading and number skills.

...

DETAILED DESCRIPTION:
This study will be the foundation of an innovative program of research designed to investigate how to communicate the complex concepts of genomics to the general public. The focus of the study will be one particular concept, the idea that genetic and environmental factors interact to affect risk of common diseases. One objective of this study will be to examine the effects of pedagogical modality (i.e., learning mode) on conceptual understanding (i.e., comprehension). A learning-by-doing (i.e., self-driven, interactive activities) condition will be compared to a learning-by-assimilation (i.e., lecture) condition to assess the effects on comprehension. The second objective of the study is to examine possible moderation of the hypothesized relationship between learning mode and comprehension by health literacy or genetic literacy (i.e., literacy skills related to these specific content areas). The third study objective is to explore possible mediators of the relationship between learning mode and comprehension. These experiments will be conducted in the NIH Immersive Virtual Environment Testing area in order to hold presentation medium constant while comparing the two learning modes. 150 participants will be for the experimental comparison phase. Because in the primary focus of the study is how the general public learns best, study participants will be healthy adult volunteers without specialized genetics knowledge. Exclusion criteria include self-reported diagnosis with epilepsy, vision or hearing problems, and vestibular disorders (e.g., dizziness, vertigo, motion sickness). Two learning-by-doing virtual environments (IVEs) and two learning-by-assimilation IVEs have been developed and pilot tested, and the IVEs that best convey the idea of gene-environment interactions have been selected for the experimental comparison. Participants will be randomized to one of two conditions: Learning-by-doing or Learning-by-assimilation; each participant will complete one IVE. The study will have two primary outcomes, both measures of comprehension: a fourteen-item measure of recall (i.e., remembering content as presented) and a six-item measure of transfer (i.e., applying content to new situations). These data will provide a foundation for a program of research investigating how best to communicate genomic concepts to the general public and, eventually, the development of effective genomic communication strategies for disease prevention interventions.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA

All participants in this study will be healthy adult volunteers. Eligibility criteria for the study are: (1) being 18-40 years of age; (2) being able to speak English and having basic English reading and writing skills; and (3) not having taken a genetics course in the past five years. Both men and women will be included in the study. We will exclude women in their last trimester of pregnancy from the study, due to the small chance of study participants tripping or bumping into walls.

Because we are interested in how members of the general public learn best about genomic topics, participants in this study will be healthy adults. Individuals who are particularly susceptible to motion sickness will be excluded. Therefore, all participants will be screened for the following conditions prior to enrollment in the study: self-reported diagnosis with epilepsy, low vision, hearing problems, or vestibular disorders (e.g., dizziness, vertigo, motion sickness).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 346
Dates: Start 2006-04-14; Primary Completion 2007-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bailenson JN, Blascovich J, Beall AC, Loomis JM. Interpersonal distance in immersive virtual environments. Pers Soc Psychol Bull. 2003 Jul;29(7):819-33. doi: 10.1177/0146167203029007002. PMID 15018671
- [Background] Baker DW, Williams MV, Parker RM, Gazmararian JA, Nurss J. Development of a brief test to measure functional health literacy. Patient Educ Couns. 1999 Sep;38(1):33-42. doi: 10.1016/s0738-3991(98)00116-5. PMID 14528569
- [Background] Collins FS, McKusick VA. Implications of the Human Genome Project for medical science. JAMA. 2001 Feb 7;285(5):540-4. doi: 10.1001/jama.285.5.540. PMID 11176855